CLINICAL TRIAL: NCT00599482
Title: Phase 1 Study to Examine the Use of Far Infrared Radiation for Pain Management During Sickle Cell Crisis
Brief Title: Far Infrared Radiation for Sickle Cell Pain Management
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GAAD Medical Research Institute Inc. (Other)
Responsible Party: Dr. Kwasi Donyina/Founder and President, GAAD Medical Research Institute Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GAAD-SCC-CTP1
Record Dates: First submitted 2008-01-11; First posted 2008-01-23 (Estimated); Last update posted 2009-01-05 (Estimated); Status verified 2009-01

CONDITIONS: Anemia, Sickle Cell
Keywords: HEMOGLOBIN SC DISEASE; HEMOGLOBIN C DISEASE; SICKLE CELL TRAIT; THALASSEMIA
MeSH Terms: conditions — Anemia, Sickle Cell; Hemoglobin SC Disease; Hemoglobin C Disease; Sickle Cell Trait; Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): Far Infrared Radiation
  Interventions: Radiation: Far Infrared Radiation (5μm to 20μm wavelength)

INTERVENTIONS:
Radiation: Far Infrared Radiation (5μm to 20μm wavelength) — Far infrared radiation for 30 to 40 minutes during each session.

SUMMARY:
Most patients with sickle-cell disease have periodic intensely painful episodes. To manage this pain, we are proposing the drinking of at least 500 mL of water followed by far infrared radiation.

DETAILED DESCRIPTION:
Painful sickle cell crises are treated with hydration and analgesics. Ischemia is an absolute or relative shortage of the blood supply to an organ. Relative shortage means the mismatch of blood supply (oxygen delivery) and blood request for adequate oxygenation of tissue.

It is hereby postulated that far infrared radiation of the body will promote blood and oxygen supply to the affected tissues. In addition, the analgesic properties of far infrared will alleviate pain due to the crisis.

ELIGIBILITY:
Inclusion Criteria:

* People with sickle cell disease

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-09 (Estimated); Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
Pain Management | 40 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ken Nedd, M.D., Study Chair — GAAD Medical Research Institute Inc.; Kwasi Donyina, Ph.D., Study Director — GAAD Medical Research Institute Inc.
Locations (1):
- The Centre for Incurable Diseases, Mississauga, Ontario, Canada